CLINICAL TRIAL: NCT00985153
Title: Comparison of the Safety, Tolerability, and Immunogenicity of 3 Consistency Lots of Frozen Measles, Mumps, Rubella, and Varicella Vaccine (ProQuad) in Healthy Children
Brief Title: Safety, Tolerability, and Immunogenicity of 3 Frozen ProQuad Consistency Lots in Healthy Children (V221-012)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V221-012; 2009_669
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2010-02-09 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ProQuad Lot 1
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 2 (Experimental): ProQuad Lot 2
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 3 (Experimental): ProQuad Lot 3
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live
- 4 (Active Comparator): M-M-R II + Varivax
  Interventions: Biological: Comparator: Varivax; Biological: Comparator: M-M-R II

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live — A Single 0.5 mL subcutaneous injection at Day 0
  Other Names: ProQuad
  Arms: 1; 2; 3
Biological: Comparator: Varivax — A Single 0.5 mL subcutaneous injection at Day 0
  Arms: 4
Biological: Comparator: M-M-R II — A Single 0.5 mL subcutaneous injection at Day 0
  Arms: 4

SUMMARY:
This study will compare three consistency lots of ProQuad to each other as well as to M-M-R II and Varivax, administered concomitantly at different injection sites, with respect to immunogenicity, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Negative clinical history of measles, mumps, rubella, varicella, and zoster

Exclusion Criteria:

* Previous receipt of measles, mumps, rubella and/or varicella vaccine either alone or in combination
* Any immune impairment or deficiency
* Exposure to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to vaccination
* Vaccination with an inactive vaccine with in the past 14 days
* Vaccination with a live vaccine within the past 30 days

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3927 (Actual)
Dates: Start 2000-03; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lieberman JM, Williams WR, Miller JM, Black S, Shinefield H, Henderson F, Marchant CD, Werzberger A, Halperin S, Hartzel J, Klopfer S, Schodel F, Kuter BJ; Consistency Lot Study Group for ProQuad. The safety and immunogenicity of a quadrivalent measles, mumps, rubella and varicella vaccine in healthy children: a study of manufacturing consistency and persistence of antibody. Pediatr Infect Dis J. 2006 Jul;25(7):615-22. doi: 10.1097/01.inf.0000220209.35074.0b. PMID 16804432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 clinical sites in the United States and 5 clinical sites in Canada
  Date of first participant visit: 12-Apr-2000
  Date of last participant visit: 11-May-2001
Groups:
- ProQuad™ Lot 1: ProQuad™ (measles, mumps, rubella, and varicella vaccine) Lot 1 administered on Day 0. ProQuad™ Lot 1 = ProQuad™ containing a varicella dose of 4.40 log10 PFU/0.5 mL.
- ProQuad™ Lot 2: ProQuad™ (measles, mumps, rubella, and varicella vaccine) Lot 2 administered on Day 0. ProQuad™ Lot 2 = ProQuad™ containing a varicella dose of 4.61 log10 PFU/0.5 mL.
- ProQuad™ Lot 3: ProQuad™ (measles, mumps, rubella, and varicella vaccine) Lot 1 administered on Day 0. ProQuad™ Lot 3 = ProQuad™ containing a varicella dose of 4.73 log10 PFU/0.5 mL.
- M-M-R™ II + VARIVAX™: VARIVAX™ + M-M-R™ II administered concomitantly at separate injection sites on Day 0.
Period: Overall Study
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Started | 985 | 968 | 962 | 1012
Vaccinated at Visit 1 | 985 | 968 | 962 | 1012
Completed | 950 | 924 | 918 | 965
Not Completed | 35 | 44 | 44 | 47
Not completed — Lost to Follow-up | 16 | 19 | 17 | 20
Not completed — Protocol Violation | 3 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 6 | 11 | 11 | 10
Not completed — Missed One or More Bleeds | 7 | 7 | 8 | 10
Not completed — Incomplete Safety Follow-up | 3 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™ | Total
Number analyzed (Participants) | 985 | 968 | 962 | 1012 | 3927
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.7 (1.3) | 12.8 (1.4) | 12.7 (1.3) | 12.8 (1.4) | 12.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478 | 448 | 442 | 468 | 1836
  Male | 507 | 520 | 520 | 544 | 2091
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 120 | 122 | 136 | 150 | 528
  Asian/Pacific | 49 | 59 | 40 | 43 | 191
  Caucasian | 615 | 630 | 622 | 647 | 2514
  Hispanic | 150 | 113 | 116 | 119 | 498
  Native American | 4 | 0 | 3 | 2 | 9
  Other | 47 | 44 | 45 | 51 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postvaccination Varicella Antibody Titer ≥ 5 Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Units/mL
Description: Antibody Response to Varicella at 6 Weeks Postvaccination for Subjects Initially With Varicella Antibody Titer < 1.25 gpELISA units/mL at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, Varicella Antibody Titer <1.25 gpELISA units/mL at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 791 | 761 | 779 | 813
Participants | 726 | 718 | 736 | 772

2. Primary Outcome: Number of Participants With Postvaccination Measles Enzyme-Linked Immunosorbent Assay (ELISA) Antibody Titer ≥ 120 mIU/mL
Description: Antibody Response to Measles at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer < 120 mIU/mL) to Measles at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 802 | 771 | 779 | 811
Participants | 790 | 753 | 753 | 800

3. Primary Outcome: Number of Participants With Postvaccination Mumps ELISA Antibody Titer ≥ 10 Ab Units/mL
Description: Antibody Response to Mumps at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer < 10 Ab units/mL) to Mumps at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 856 | 823 | 830 | 872
Participants | 825 | 796 | 788 | 854

4. Primary Outcome: Number of Participants With Postvaccination Rubella ELISA Antibody Titer ≥ 10 IU/mL
Description: Antibody Response to Rubella at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer < 10 IU/mL) to Rubella at Baseline
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 861 | 835 | 836 | 866
Participants | 852 | 821 | 828 | 859

5. Primary Outcome: Antibody Response to Varicella for Subjects Initially With Varicella Antibody Titer < 1.25 gpELISA Units/mL at Baseline - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Varicella
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, Varicella Antibody Titer < 1.25 gpELISA units/mL at baseline, and followed protocol procedures.
Measure: Mean (95% Confidence Interval); unit: gpELISA
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 791 | 761 | 779 | 813
gpELISA | 16.0 [14.9 to 17.2] | 18.4 [17.2 to 19.7] | 19.7 [18.4 to 21.0] | 17.6 [16.6 to 18.7]

6. Primary Outcome: Antibody Response to Measles for Subjects Initially Seronegative (a Titer < 120 mIU/mL) to Measles at Baseline - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Measles.
Time Frame: 6 weeks Postvaccination
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 802 | 771 | 779 | 811
mIU/mL | 3031.6 [2841.6 to 3234.3] | 2939.3 [2740.0 to 3153.2] | 2852.2 [2651.0 to 3068.7] | 2095.6 [1964.2 to 2235.7]

7. Primary Outcome: Antibody Response to Mumps for Subjects Initially Seronegative (a Titer < 10 Ab Units/mL) to Mumps at Baseline - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Mumps.
Time Frame: 6 weeks Postvaccination
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ELISA AB units
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 856 | 823 | 830 | 872
ELISA AB units | 100.5 [94.3 to 107.2] | 102.3 [96.0 to 109.0] | 85.6 [79.9 to 91.8] | 89.7 [84.7 to 94.9]

8. Primary Outcome: Antibody Response to Rubella for Subjects Initially Seronegative (a Titer < 10 IU/mL) to Rubella at Baseline - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to Rubella
Time Frame: 6 weeks Postvaccination
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ELISA AB units
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 861 | 835 | 836 | 866
ELISA AB units | 113.5 [107.5 to 119.8] | 114.8 [108.2 to 121.8] | 114.2 [108.1 to 120.6] | 132.6 [125.7 to 140.0]

9. Primary Outcome: Number of Participants With Serious Vaccine-related CAEs
Description: Subjects with a serious vaccine-related CAE (an AE which is assessed by an investigator/qualified physician as being related to study vaccine and results in death, persistent or significant disability/incapacity, prolongs an existing inpatient hospitalization, is life-threatening, a congenital anomaly/birth defect, a cancer, or an overdose).
Time Frame: 6 weeks Postvaccination
Population: All subjects with follow-up for safety were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Number analyzed (Participants) | 969 | 950 | 941 | 993
Participants
  With Serious Vaccine-Related CAEs | 2 | 1 | 2 | 1
  Without Serious Vaccine-Related CAEs | 967 | 949 | 939 | 992

ADVERSE EVENTS:
Description: Number of participants reported as "At Risk" is the number of participants with follow-up.
Arm/Group | ProQuad™ Lot 1 | ProQuad™ Lot 2 | ProQuad™ Lot 3 | M-M-R™ II + VARIVAX™
Serious Adverse Events (participants affected / at risk) | 6/969 | 8/950 | 11/941 | 11/993
Other Adverse Events (participants affected / at risk) | 793/969 | 758/950 | 769/941 | 785/993
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProQuad™ Lot 1 (N=969) | ProQuad™ Lot 2 (N=950) | ProQuad™ Lot 3 (N=941) | M-M-R™ II + VARIVAX™ (N=993)
Seizure, febrile (Nervous system disorders) | 2 | 1 | 2 | 3
Seizure disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Accidental ingestion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 2 | 1
Infection, urinary tract (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Otitis media (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Fracture, humerus, right (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fracture, radius, right (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Infection, RSV (Infections and infestations) | 0 | 1 | 1 | 0 — Infection, respiratory syncytial virus (RSV)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Gastroenteritis, Infectious (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infection, viral (Infections and infestations) | 0 | 0 | 2 | 0
Hypovolemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Bite, animal (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pyelonephritis (General disorders) | 0 | 0 | 1 | 0
Drug abuse (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 — Drug abuse refers to cocaine metabolites found in subject's urine.
Allergy (Immune system disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Breathing Pattern Abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ProQuad™ Lot 1 (N=969) | ProQuad™ Lot 2 (N=950) | ProQuad™ Lot 3 (N=941) | M-M-R™ II + VARIVAX™ (N=993)
Fever (General disorders) | 379 | 362 | 378 | 327
Infection, Viral (Infections and infestations) | 41 | 29 | 30 | 30
Trauma (Injury, poisoning and procedural complications) | 10 | 11 | 10 | 6
Anorexia (Metabolism and nutrition disorders) | 18 | 21 | 18 | 20
Constipation (Gastrointestinal disorders) | 7 | 9 | 10 | 12
Diarrhea (Gastrointestinal disorders) | 80 | 80 | 77 | 81
Gastroenteritis (Gastrointestinal disorders) | 18 | 30 | 21 | 20
Gastroenteritis, Infectious (Infections and infestations) | 13 | 5 | 8 | 15
Vomiting (Gastrointestinal disorders) | 59 | 48 | 58 | 60
Irritability (Psychiatric disorders) | 105 | 101 | 119 | 86
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 16 | 9
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 6 | 7
Congestion, Nasal (Respiratory, thoracic and mediastinal disorders) | 15 | 10 | 14 | 18
Congestion, Respiratory (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 18 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 57 | 55 | 61 | 61
Infection, Respiratory, Upper (Infections and infestations) | 280 | 248 | 249 | 245
Influenza (Infections and infestations) | 10 | 9 | 10 | 8
Laryngotracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 10 | 14
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 25 | 15 | 29 | 21
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 58 | 65 | 58 | 60
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 18 | 14 | 8 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 9 | 14
Bite/Sting, Non-Venomous (Injury, poisoning and procedural complications) | 7 | 7 | 15 | 12
Dermatitis, Contact (Skin and subcutaneous tissue disorders) | 20 | 15 | 20 | 21
Eczema (Skin and subcutaneous tissue disorders) | 18 | 19 | 14 | 19
Laceration (Skin and subcutaneous tissue disorders) | 4 | 5 | 7 | 10
Miliaria Rubra (Skin and subcutaneous tissue disorders) | 16 | 24 | 23 | 22
Rash (Skin and subcutaneous tissue disorders) | 59 | 51 | 54 | 45
Rash, Diaper (Skin and subcutaneous tissue disorders) | 72 | 78 | 80 | 86
Rash, Measles/Rubella-Like (Skin and subcutaneous tissue disorders) | 30 | 24 | 24 | 19
Rash, Varicella-Like (Skin and subcutaneous tissue disorders) | 30 | 18 | 15 | 24
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 15 | 2 | 10
Viral Exanthema (Infections and infestations) | 54 | 41 | 47 | 45
Conjunctivitis (Eye disorders) | 27 | 12 | 25 | 21
Otitis (Ear and labyrinth disorders) | 30 | 27 | 17 | 18
Otitis Media (Ear and labyrinth disorders) | 133 | 109 | 133 | 117
Ecchymosis (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 17 | 14 | 16 | 0/0
Erythema (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 149 | 163 | 163 | 0/0
Pain/Tenderness/Soreness (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 221 | 246 | 230 | 0/0
Rash (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 13 | 33 | 35 | 0/0
Swelling (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 89 | 86 | 86 | 0/0
Ecchymosis (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 15
Erythema (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 136
Pain/Tenderness/Soreness (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 262
Rash (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 17
Swelling (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 91
Ecchymosis (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 15
Erythema (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 134
Pain/Tenderness/Soreness (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 266
Swelling (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 80

LIMITATIONS AND CAVEATS:
One additional subject received M-M-R™ II and ProQuad™ vaccines at the same visit in error; this child was excluded from all immunogenicity and safety summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.